CLINICAL TRIAL: NCT00693433
Title: A Phase 1 Study of CCI-779 in Combination With Dexamethasone in Multiple Myeloma
Brief Title: Temsirolimus and Dexamethasone in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00157; VAMC-SC-7353; CDR0000597181
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-06

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; temsirolimus; Sirolimus

ARMS (1):
- Treatment (enzyme inhibitor, chemotherapy) (Experimental): Patients receive temsirolimus IV over 30 minutes once weekly on days 1, 8, 15, and 22 and oral dexamethasone once on days 1, 2, 8, 9, 15, 16, 22, and 23. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dexamethasone; Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given together with dexamethasone in treating patients with recurrent or refractory multiple myeloma. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus together with dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity and safety of temsirolimus in combination with dexamethasone in patients with recurrent or refractory multiple myeloma.

II. To assess a dose of temsirolimus that is capable of inhibiting the mammalian target of rapamycin (mTOR) in myeloma tumor cells.

SECONDARY OBJECTIVES:

I. To assess the efficacy of temsirolimus in combination with dexamethasone in these patients.

II. To correlate the efficacy of this regimen with molecular characteristics of the individual tumor clones.

OUTLINE: This is a multicenter, dose-escalation study of temsirolimus.

Patients receive temsirolimus intravenously (IV) over 30 minutes once weekly on days 1, 8, 15, and 22 and oral dexamethasone once on days 1, 2, 8, 9, 15, 16, 22, and 23. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow aspiration and blood sample collection periodically for correlative studies. Correlative studies include analysis of p70S6 kinase activity in peripheral blood mononuclear cells and in multiple myeloma cells; analysis of the degree of AKT phosphorylation and degree of PTEN expression in multiple myeloma cells by immunohistochemistry; Ras mutational analysis; and Myc 5'UTR mutational analysis.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed multiple myeloma

  * Measurable levels of M protein in serum and/or urine
* Recurrent or refractory disease

  * Progressive disease after treatment with ≥ 2 separate chemotherapeutic regimens

    * At least 1 of the regimens must have included high-dose dexamethasone (40 mg on days 1-4, 9-12, and 17-20) or medium-dose dexamethasone (40 mg on days 1, 8, 15, and 22) of a 28-day course
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm ^3
* Total bilirubin < 2 mg/dL
* AST and ALT < 3 times upper limit of normal
* Creatinine < 2 mg/dL
* Fasting cholesterol < 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to temsirolimus or dexamethasone
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Poorly controlled hypertension
  * Diabetes mellitus
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* See Disease Characteristics
* At least 4 weeks since prior cytotoxic therapy
* More than 4 weeks since prior chemotherapy and recovered
* No concurrent anticonvulsive or antiarrhythmic medications
* No concurrent enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital) or other CYP3A4 inhibitors or inducers (e.g., rifampin or Hypericum perforatum [St. John wort])
* No concurrent prophylactic hematopoietic colony-stimulating factors
* No other concurrent investigational therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of temsirolimus | Course 1 (first 28 days)
  The MTD is the dose level at which less than 2 out of 6 subjects experience DLT. Assessed according to the NCI Common Toxicity Criteria (CTC).
Toxicity and safety | Continuously from start of treatment study
  The description and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for AE reporting.

SECONDARY OUTCOMES:
Correlation between response to treatment with temsirolimus and the degree of p70 inhibition in peripheral blood mononuclear cells and in multiple myeloma (MM) cells | Every 4 weeks
  We will examine a scatter plot of the absolute and Percent change in PBMNC versus the absolute and percent change in BM. Spearman (non-parametric) and Pearson (parametric) correlation coefficients and linear and/or spline smoothing regression on either the original or a transformed scale will be used to assess the relationship. We will compare mean and median levels in those who respond versus those who do not using the Wilcoxon rank sum test and we will report the percent of overlap in P70 between the two groups. Assessed using analysis of variance methods or their non-parametric analog.
Correlation between response to treatment with temsirolimus and the degree of pre-treatment AKT activation in MM cells | Every 4 weeks
  Assessed by immunohistochemistry (IHC). We will first carry out a bivariate assessment of AKT percent positivity versus the binary outcome of response versus no response to treatment. For AKT score, we will compare mean and median levels in those who respond versus those who do not using the Wilcoxon rank sum test and we will report the percent of overlap in AKT between the two groups.
Correlation between response to treatment with temsirolimus and the degree of PTEN expression in MM cells | Every 4 weeks
  PTEN expression will be determined by IHC. We will first carry out a bivariate assessment of PTEN score versus the binary outcome of response versus no response to treatment. For PTEN variables, we will report the corresponding contingency table versus response and use Wilcoxon test to assess the association if applicable.
Correlation between response to treatment with temsirolimus and the presence of RAS mutations | Every 4 weeks
  We will first carry out a bivariate assessment of RAS mutational status versus the binary outcome of response versus no response to treatment. For RAS variables, we will report the corresponding contingency table versus response and use Fishers exact test to assess the association.
Correlation between response to treatment with temsirolimus and the presence of myc mutations | Every 4 weeks
  We will first carry out a bivariate assessment of MYC mutational status versus the binary outcome of response versus no response to treatment. For MYC variables, we will report the corresponding contingency table versus response and use Fishers exact test to assess the association.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lichtenstein, Principal Investigator — Veterans Administration Los Angeles Healthcare System
Locations (1):
- Veteran's Administration Medical Center, Las Angeles, California, United States